CLINICAL TRIAL: NCT05088850
Title: The Early Prediction of Sepsis Occurrence in ICU
Brief Title: The Early Prediction of Sepsis in ICU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, lei li, chief physician, Ruijin Hospital
Other Study IDs: 20211014LILEI
Record Dates: First submitted 2021-10-18; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Prediction of Sepsis in Critical Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-sepsis
  Interventions: Other: no intervention
- sepsis
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Sepsis is a vital issue in critical care medicine, and early detection and intervention are key to survival. We aimed to establish an early warning system for sepsis based on a data integration platform that can be implemented in the ICU.

ELIGIBILITY:
Inclusion Criteria:

Patients who met all of the following criteria were included in the case group:

1. At least 14 years old.
2. Sepsis onset at least 5 hours after ICU admission.
3. Sepsis onset is the first instance since admission to the hospital.

Exclusion Criteria:

Patients meeting all of the following criteria were included in the control group:

1. At least 14 years old.
2. Patients staying in ICU for at least 5 hours and have not had sepsis in this time.
3. Patients without ICD-9 codes for sepsis (785·52, 995·91, 995·92).
4. SOFA score change is not more than 1 point in an arbitrary continuous 72 hours in the ICU stay.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients that were admitted into the ICU.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-05-30 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
confidence index of sepsis occurrence | sepsis occurrence in five hours

CONTACTS AND LOCATIONS:
Locations (1):
- ICU, Ruijin Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Chen Q, Li R, Lin C, Lai C, Chen D, Qu H, Huang Y, Lu W, Tang Y, Li L. Transferability and interpretability of the sepsis prediction models in the intensive care unit. BMC Med Inform Decis Mak. 2022 Dec 29;22(1):343. doi: 10.1186/s12911-022-02090-3. PMID 36581881